CLINICAL TRIAL: NCT07393360
Title: Evaluating the Effect of a Food for Special Medical Purposes Containing Essential Amino Acids (EAA), Carnitine, Arginine, and Sucrosomial Minerals on the Preservation of Appendicular Skeletal Muscle Mass (ASMM) During a Weight Loss Program With GLP-1 Receptor Agonists
Brief Title: Effect of a Food for Special Medical Purposes on Muscle Mass Preservation During GLP-1 RAs Weight Loss Treatment
Acronym: MYO-PRESERVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanutra S.p.a. (Industry)
Collaborators: Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MYO-PRESERVE
Record Dates: First submitted 2025-12-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight
Keywords: Weight Loss; Muscle Mass Preservation; Obesity; Body Composition; BIVA
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active product and placebo are indistinguishable in appearance, packaging, and administration schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myosave® (Experimental): Participants receive Myosave® twice daily (two sachets/day) for 24 weeks, in addition to standard GLP-1 RA or dual GIP/GLP-1 RA therapy.
  Interventions: Dietary Supplement: Myosave®
- Placebo (Placebo Comparator): Participants receive a matching placebo twice daily for 24 weeks, in addition to standard GLP-1 RA or dual GIP/GLP-1 RA therapy.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Myosave® — A Food for Special Medical Purposes. Two sachets per day (morning and afternoon), taken on an empty stomach for 24 weeks.
  Arms: Myosave®
Other: Placebo — Maching in appearance, taste, and dosing schedule to Myosave®. Two sachets per day for 24 weeks
  Arms: Placebo

SUMMARY:
This study evaluates whether a Food for Special Medical Purposes (FSMP) can help to preserve appendicular skeletal muscle mass (ASMM) in adults undergoing weight loss treatment with GLP-1 receptor agonists or dual GIP/GLP-1 receptor agonists. Participants will receive the FSMP or a matching placebo for 24 weeks while continuing standard GLP-1-based therapy. ASMM will be measured using Bioelectrical Impedance Vector Analysis (BIVA).

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled investigates whether a Food for Special Medical Purposes (FSMP) can help preserve appendicular skeletal muscle mass (ASMM) in adults undergoing weight loss treatment with GLP-1 receptor agonists or dual GIP/GLP-1 receptor agonists.

Eligible participants are adults with obesity or overweight with comorbidities who are initiating GLP-1-based therapy as part of standard clinical management. Participants are randomized in a 1:1 ratio to receive either the FSMP or a matching placebo for 24 weeks, in addition to their ongoing GLP-1 RA or dual GIP/GLP-1 RA therapy. Study visits occur at baseline, 8 weeks, 16 weeks, and 24 weeks.

This trial aims to determine whether targeted nutritional support can mitigate the loss of lean mass commonly observed during pharmacologically assisted weight loss, thereby improving functional outcomes and overall patient well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤ 65 years old;
* BMI ≥ 30 Kg/m2 and ≤45 kg/m2
* BMI from 27 kg/m2 to 30 Kg/m2 with at least one associated co-morbidity related to overweight [e.g. dysglycemia (pre-diabetes and/or metabolic syndrome), hypertension, dyslipidemia, obstructive sleep apnea syndrome (OSAS], or cardiovascular disease]
* Starting to use a GLP-1 RAs (liraglutide, semaglutide) or dual GIP and GLP-1 RAs (tirzepatide) for weight reduction; patient can be enrolled if they start the treatment at the time of enrollment or up to 2 weeks
* Diet composition adjusted to provide 0.9-1.1 g/Kg ideal body weight proteins
* Signed informed consent

Exclusion Criteria:

* Type I and Type II diabetes; patients with pre-diabetes and/or metabolic syndrome and assuming Metformin and SGLT-2 inhibitors can be enrolled
* Monogenic obesity (Subjects with a known diagnosis of monogenic obesity, including but not limited to pathogenic mutations in LEP, LEPR, MC4R, POMC, PCSK1, or other genes known to cause monogenic forms of early-onset or syndromic obesity)
* Reduced kidney function, defined as eGFR < 60 mL/min/1.73 m², calculated using the CKD-EPI equation (see Appendix 1)
* Oncologic patients in active treatments
* Hypersensitivity to any of the constituents of the study product
* Pregnancy
* Breastfeeding
* Use of meal replacements for a diet enriched with aminoacids and/or HMB
* Use of food supplements containing aminoacids and/or HMB; patients can be included in the study if they undergo a washout period of at least 15 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Appendicular Skeletal Muscle Mass (ASMM) | Baseline, Week 8, Week 16, Week 24
  ASMM will be assessed using Bioelectrical Impedance Vector Analysis (BIVA). The primary endpoint is the change in ASMM from baseline to Week 24 to determine whether the Food for Special Medical Purposes (FSMP) preserves skeletal muscle mass compared with placebo.

SECONDARY OUTCOMES:
Handgrip Strength | Baseline, Week 8, Week 16, Week 24
  Handgrip strength will be measured with a calibrated dynamometer on both dominant and non-dominant hands to evaluate changes in muscle function.
Change in Fat-Free Mass (FFM) | Baseline, Week 8, Week 16, Week 24
  Change in Fat-Free Mass measured using Bioelectrical Impedance Vector Analysis (BIVA). Continuous variable reported according to device output.
Change in Fat Mass (FM) | Baseline, Week 8, Week 16, Week 24
  Change in Fat Mass measured using Bioelectrical Impedance Vector Analysis (BIVA). Continuous variable reported according to device output.
Change in Health-Related Quality of Life (Short Form-36 Health Survey, SF-36) | Baseline, Week 8, Week 16, Week 24
  The Short Form-36 Health Survey (SF-36) assesses physical and mental health-related quality of life.
  The scale consists of 36 items scored into 8 domains. Each domain score ranges from 0 to 100, where higher scores indicate better health status.
  Domains include: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health.
Change in Body Weight (kg) | Baseline to Week 24
  Change in body weight measured in kilograms from baseline to Week 24. Continuous variable reported according to standard clinical procedures.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS Auxologico, Milan
  - IRCCS San Raffaele, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano